CLINICAL TRIAL: NCT04067648
Title: Effect of Three Doses of Sufentanil on Anesthesia Introduction and Recovery Quality in Pediatric Adenotonsillectomy
Brief Title: Sufentanil on Anesthesia Introduction and Recovery Quality in Pediatric Adenotonsillectomy
Acronym: SFTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, associate professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFTA
Record Dates: First submitted 2019-08-17; First posted 2019-08-26 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Sufentanil
Keywords: Sufentanil; perfusion index
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Observers and patients were double-blind. Sufentanil was assigned by a specialist. Different doses of sufentanil were allocated in the same volume according to the weight of the child.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- S1 group (Experimental): Sufentanil 0.3 μg/kg was intravenously given during anesthesia induction
  Interventions: Drug: Sufentanil Injection
- S2 group (Experimental): Sufentanil 0.4 μg/kg was intravenously given during anesthesia induction
  Interventions: Drug: Sufentanil Injection
- S3 group (Experimental): Sufentanil 0.5 μg/kg was intravenously given during anesthesia induction
  Interventions: Drug: Sufentanil Injection

INTERVENTIONS:
Drug: Sufentanil Injection — three doses of sufentanil was intravenously given during anesthesia induction
  Other Names: adenotonsillectomy

SUMMARY:
To study the effect of different doses of sufentanil on anesthesia induction and analgesia after tonsillectomy in children. According to the different doses of sufentanil used in anesthesia induction, the children were divided into 3groups. The vital signs during anesthesia, the recovery period of anesthesia and the complications after anesthesia were compared among the groups. The anesthetic effects and safety of sufentanil at different doses were discussed, which provided theoretical basis for clinical selection of the best drug dosage.

DETAILED DESCRIPTION:
Fifteen minutes before operation, midazolam 0.1 mg/kg was slowly intravenously injected. Five minutes later, the child entered the operating room. Pi, Narcotrend, blood pressure, ECG, SpO2 and body temperature were monitored. Penehyclidine hydrochloride 0.01 mg/kg, dexamethasone 0.1 mg/kg, propofol 3 mg/kg, sufentanil (0.3μg/kg, 0.4 μg/kg, 0.5 μg/kg) were given during anesthesia induction. cis-atracurium 0.15 mg/kg, using the required type of tube for tracheal intubation. Sevoflurane 1.0 MAC + remifentanil 0.15 ug/kg/min 50% oxygen was given during anesthesia maintenance. Effective analgesia was achieved by adjusting the dosage of remifentanil during operation.

The changes of vital signs including perfusion index, Narcotrend, Bp, HR, oxygen saturation were observed before anesthesia induction, immediately after tracheal intubation, during tonsillectomy and adenoidectomy during operation, after extubation and in the recovery room. Then record the recovery time, restlessness and pain score during recovery period, postoperative pain, nausea and vomiting and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-12 years,
* ASA I-II grade;
* selective adenotonsillectomy
* BMI 18.5～23.9,
* Sign informed consent

Exclusion Criteria:

* Emergency surgery;
* Abnormal liver and kidney function
* severe dehydration and malnutrition or Hb < 10g/dl;
* BMI <18.5 or <23.9;
* Children with neurological disorders

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
adequate sufentanil dose | 24 hours
  Adequate sufentanil dose is determined by Optimal intubation conditions and No hypotension or other severe side effects

SECONDARY OUTCOMES:
cut off value of Pi for valid stress assessment | 24 hours
  a validated and useful stress assessment for children during endotracheal intubation.
Narcotrend index | 24 hours
  explore dose and age-related hemodynamic effects of sufentanil. Next to blood pressure and heart rate and continuous Narcotrend will be monitored. Then record the correlation between perfusion index and Narcotrend
postoperative complications with different doses of sufentanil | 7days
  Including postoperative pain and the dosage of analgesics after operation and the satisfaction of children and parents

CONTACTS AND LOCATIONS:
Overall Officials: Aijun XU, Dr., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
According to the results of the experiment and the opinions of the children's families, it is decided whether to publish the data or not.